CLINICAL TRIAL: NCT00409682
Title: A Multi-Center, Double-Blind Study to Evaluate the Safety, Efficacy and Pharmacokinetics of the Human Anti-TNF Monoclonal Antibody Adalimumab in Pediatric Subjects With Moderate to Severe Crohn's Disease
Brief Title: Efficacy and Safety of Adalimumab in Pediatric Subjects With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Andreas Lazar, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-806; 2006-004814-41 (EudraCT Number)
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open-label adalimumab (Week 0 to Week 4) (Active Comparator): All subjects received an open-label adalimumab induction regimen. Subjects weighing greater than or equal to 40 kg at Baseline received 160 mg at Week 0 and 80 mg at Week 2. Subjects weighing less than 40 kg at Baseline received 80 mg at Week 0 and 40mg at Week 2.
  Interventions: Biological: Adalimumab
- Low-Dose Adalimumab: 20 mg or 10 mg eow (Week 4 to Week 52) (Active Comparator): Subjects randomized to the Low-Dose treatment group received either 20 mg adalimumab every other week (eow) (if Week 4 body weight [BW] was greater than or equal to 40 kg) or 10 mg adalimumab eow (if Week 4 BW less than 40 kg). Starting at the Week 12 study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blind (DB) ew therapy they could be switched to open-label ew therapy.
  Interventions: Biological: Adalimumab
- High-Dose Adalimumab: 40 mg or 20 mg eow (Week 4 to Week 52) (Active Comparator): Subjects randomized to the High-Dose treatment group received either 40 mg adalimumab every other week (eow) (if Week 4 body weight [BW] was greater than or equal to 40 kg) or 20 mg adalimumab eow (if Week 4 BW less than 40 kg). Starting at the Week 12 study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blinded (DB) ew therapy they could be switched to open-label ew therapy.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — All subjects received an open-label adalimumab induction regimen. Subjects weighing greater than or equal to 40 kg at Baseline received 160 mg at Week 0 and 80 mg at Week 2. Subjects weighing less than 40 kg at Baseline received 80 mg at Week 0 and 40mg at Week 2.
  Other Names: ABT-D2E7, adalimumab, Humira
  Arms: Open-label adalimumab (Week 0 to Week 4)
Biological: Adalimumab — Subjects randomized to the Low-Dose treatment group received either 20 mg adalimumab every other week (eow) (if Week 4 body weight [BW] was greater than or equal to 40 kg) or 10 mg adalimumab eow (if Week 4 BW less than 40 kg). Starting at the Week 12 study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blind (DB) ew therapy they could be switched to open-label ew therapy.
  Other Names: ABT-D2E7, adalimumab, Humira
  Arms: Low-Dose Adalimumab: 20 mg or 10 mg eow (Week 4 to Week 52)
Biological: Adalimumab — Subjects randomized to the High-Dose treatment group received either 40 mg adalimumab every other week (eow) (if Week 4 body weight [BW] was greater than or equal to 40 kg) or 20 mg adalimumab eow (if Week 4 BW less than 40 kg). Starting at the Week 12 study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blinded (DB) ew therapy they could be switched to open-label ew therapy.
  Other Names: ABT-D2E7, adalimumab, Humira
  Arms: High-Dose Adalimumab: 40 mg or 20 mg eow (Week 4 to Week 52)

SUMMARY:
The purpose of this study is to determine Efficacy, Pharmacokinetics, and Safety of Adalimumab in Pediatric Subjects With Moderate to Severe Crohn's Disease

DETAILED DESCRIPTION:
M06-806 (NCT # NCT00409682) was a Phase 3, multi-center, randomized, double-blind (DB), efficacy, safety, and pharmacokinetic (PK) study designed to evaluate the efficacy of 2 dose regimens for the induction and maintenance of clinical remission in pediatric subjects between the ages of 6 and 17 (inclusive) with moderate to severe Crohn's disease (CD) (defined by Pediatric Crohn's Disease Activity Index [PCDAI > 30]). Subjects must have either failed conventional therapy for CD or have previously received infliximab and lost response/had intolerance to infliximab.

Approximately 186 pediatric subjects between the ages of 6 and 17 were planned to be entered into the study at approximately 55 sites in the US, Canada, and Europe. At least 80 subjects were to be ≥ 13 years old at Baseline and one-third to one-half of the study population were to be subjects who had previously lost response or were intolerant to infliximab.

The duration of the study was to be up to 65 weeks, which included a 1- to 3-week Screening period, an Induction period, a Maintenance period, and a 70-day follow-up phone call for all subjects that either terminated early from the study or did not rollover into the extension study ([NCT # 00686374], to evaluate the long-term maintenance of clinical response, safety, and tolerability of repeated administration of adalimumab).

All subjects received an induction regimen administered at Baseline (Week 0) and Week 2. The open-label (OL) induction dose was based on the subject's Baseline body weight. Subjects weighing ≥ 40 kg were to receive 160 mg at Week 0 and 80 mg adalimumab at Week 2. Subjects weighing < 40 kg were to receive 80 mg at Week 0 and 40 mg adalimumab at Week 2.

At Week 4, subjects were to be randomized 1:1 to 1 of 2 DB maintenance treatment groups (Low-Dose or High-Dose), stratified by Week 4 clinical responder status (clinical response was defined as decrease in PCDAI of ≥ 15 points from the Baseline score), body weight at Week 4 and prior exposure to infliximab. Subjects randomized to the High-Dose treatment group were to receive either 40 mg adalimumab subcutaneous (SC) every other week (eow) (if Week 4 body weight ≥ 40 kg) or 20 mg adalimumab SC eow (if Week 4 body weight < 40 kg). Subjects randomized to the Low-Dose treatment group were to receive either 20 mg adalimumab SC eow (if Week 4 body weight ≥ 40 kg) or 10 mg adalimumab SC eow (if Week 4 body weight < 40 kg).

Subject's body weight taken at Week 26 was to be used to readjust the maintenance dosing regimen for a subject whose body weight had increased from < 40 kg to ≥ 40 kg during the study.

Subjects were expected to remain on blinded eow therapy throughout the 48-week study DB Maintenance period. However, starting at the Week 12 study visit, subjects who experienced a disease flare (increase in the PCDAI ≥ 15 points when compared to Week 4 and an absolute PCDAI above 30) or were non-responders (not achieving a decrease in the PCDAI score of at least 15 points when compared to the Baseline score for 2 consecutive visits at least 2 weeks apart) could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. During blinded ew treatment, if a subject continued to experience a flare or met the definition of non-response following an 8 week course of DB ew therapy, they were to be switched to OL ew therapy. The dosage of the OL ew therapy was 20 mg for subjects < 40 kg and 40 mg for subjects ≥ 40 kg.

This study used the PCDAI to determine efficacy of the study drug. The primary efficacy endpoint is the proportion of subjects who are in clinical remission at Week 26, as measured by the PCDAI in the intent-to-treat population. Clinical remission is defined as a PCDAI score of ≤ 10.

The clinical response indicators include clinical remission as defined by PCDAI score at Week 52 and clinical response as defined by PCDAI score at Week 26 and at Week 52.

The patient reported outcome is the change from Baseline in total IMPACT III scores at Week 26 and Week 52.

The safety parameters (adverse events, laboratory data, and vital signs) were assessed at all visits throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 6 and 17, inclusive, prior to baseline dosing.
2. Subjects with a diagnosis of Crohn's disease for greater than 12 weeks prior to screening, confirmed by endoscopy or radiologic evaluation.
3. PCDAI > 30 despite concurrent treatment with an oral corticosteroid, and/or azathioprine (AZA) or 6-mercaptopurine (6-MP) or methotrexate (MTX) as defined below:

   * Oral corticosteroid - Prednisone of ≥ 10 mg/day or equivalent, but not exceeding 40 mg, with a stable dose for at least two weeks prior to Baseline.
   * Azathioprine or 6-MP - AZA dose of ≥ 1.5 mg/kg/day or 6-MP dose of ≥ 1 mg/kg/day rounded to the nearest available tablet formulation, or a dose that is the highest tolerated for the subject, in the opinion of the investigator (for example due to leukopenia, elevated liver enzymes, nausea, etc.) for at least 8 weeks prior to Baseline with a stable dose for at least 4 weeks prior to Baseline.
   * MTX dose of ≥ 5 mg once weekly, either subcutaneously (SC), intramuscularly (IM), or orally for subjects whose body weight is ≥ 20 kg, or a dose that is the highest tolerated for the subject, in the opinion of the investigator (for example due to leukopenia, elevated liver enzymes, nausea, etc.) for at least 8 weeks prior to Baseline with a stable dose for at least 4 weeks prior to Baseline.
   * MTX dose of 0.2 mg/kg, up to 5 mg, once weekly, either SC, IM, or orally for subjects whose body weight is < 20 kg, or a dose that is the highest tolerated for the subject, in the opinion of the investigator (for example due to leukopenia, elevated liver enzymes, nausea, etc.) for at least 8 weeks prior to Baseline with a stable dose for at least 4 weeks prior to Baseline.
   * Concurrent therapy will not be required for subjects who within the past 2 years in the opinion of the Investigator have not responded to or could not tolerate systemic corticosteroids, AZA, 6-MP, or MTX as defined below:

     * Corticosteroids:

       * Failed to successfully respond to corticosteroids, or
       * Medical complications and/or adverse events (AEs) from corticosteroids that in the judgment of their physician, precludes their use (e.g. psychosis, uncontrolled diabetes, osteoporosis, or osteonecrosis).
     * Azathioprine, 6-MP or MTX: -

       * Failed to successfully respond to these drugs or
       * Medical complications and/or AEs that in the judgment of their physician, precludes their use (e.g. allergic reaction, pancreatitis, elevated liver enzymes, hepatitis or leukopenia).
4. If female, subjects who were sexually active and were of child-bearing potential practicing an approved method of birth control throughout the study and for 150 days after study completion. Examples of approved methods of birth control included the following:

   * Condoms, sponge,foam,jellies,diaphragm, or intrauterine device (IUD)
   * Oral,parenteral, or intravaginal contraceptives for 12 weeks prior to adalimumab administration
   * A vasectomized partner.
5. Parent or legal guardian,as required,had voluntarily signed and dated an informed consent form (IFC), approved by an Institutional Review Board (IRB)/ Independent Ethics Committee (IEC).
6. Adequate cardiac, renal and hepatic function as determined by principal investigator and demonstrated by Screening laboratory evaluations, questionnaires, and physical examination results that are within normal limits.
7. Parent or legal guardian was willing to actively supervise storage and administration of study drug and to ensure that the time of each dose was accurately recorded in the subject's diary.
8. Subjects who had previously received infliximab, providing the subject had an initial response and then discontinued use due to a loss of response, or discontinued use due to intolerance.

Exclusion Criteria:

1. History of cancer or lymphoproliferative disease other than a successfully and completely treated cutaneous squamous cell or basal cell carcinoma or carcinoma-in-situ of the cervix.
2. History of listeria, histoplasmosis, chronic or active hepatitis B infection, human immunodeficiency virus (HIV), an immunodeficiency syndrome, central nervous system (CNS) demyelinating disease, or active tuberculosis (TB) (receiving treatment or not receiving treatment), severe infections such as sepsis and opportunistic infections.
3. Subject with infectious colitis, ulcerative colitis or indeterminate colitis as determined by the investigator and Abbott Medical Monitor.
4. Subject with symptomatic known obstructive strictures.
5. Subject who had surgical bowel resections within the past 24 weeks of the Baseline visit or planned any resection at any time point while enrolled in the study.
6. Subject with an ostomy or ileo-anal pouch. (Subjects with a previous ileo-rectal anastomosis were not excluded).
7. Subject who had short bowel syndrome as determined by the investigator.
8. Subject who was currently receiving total parenteral nutrition (TPN).
9. Females who were pregnant or were currently breast-feeding.
10. Subject who had received any investigational chemical agent in the past 30 days or 5 half-lives prior to Baseline (whichever was longer).
11. Subject who had received any investigational biological agent in the past 16 weeks or 5 half-lives prior to Baseline (whichever was longer).
12. Subject who has had systemic antibiotic, antiviral or antifungal treatment(s) within 3 weeks prior to Baseline for any non-Crohn's related infections.
13. Subject with a history of clinically significant drug or alcohol abuse in the last year.
14. Subjects with a poorly controlled medical condition such as: uncontrolled diabetes, recurrent infections, unstable ischemic heart disease, moderate to severe heart failure, recent cerebrovascular accidents and any other condition which, in the opinion of the investigator or the Sponsor, would put the subject at risk by participation in the protocol.
15. Subjects with positive C. difficile stool assay.
16. Subject who previously used infliximab within eight weeks of Baseline.
17. Subject who previously used infliximab and had not clinically responded at any time ("primary non-responder") unless subject experienced a treatment limiting reaction to infliximab.
18. Previous treatment with any other anti-TNF agent except infliximab.
19. Received previous treatment with adalimumab or previous participation in an adalimumab clinical study.
20. Screening laboratory and other analyses showing any of the following abnormal results:

    * Electrocardiogram (ECG) - with clinically significant abnormalities;
    * Aspartate transaminase (AST) or alanine transaminase (ALT) >1.75 x the upper limit of the reference range;
    * Total bilirubin ≥ 3 mg/dL;
    * Serum creatinine > 1.6 mg/dL;
21. Subjects on AZA, 6-MP, or MTX who had not been on these medications for at least 8 weeks prior to Baseline and on stable doses of these medications for at least 4 weeks prior to Baseline. Subjects who had been on AZA, 6-MP, or MTX who had discontinued these medications within 8 weeks of Baseline.
22. Subjects on aminosalicylates, or Crohn's-related antibiotics (fluoroquinolones such as ciprofloxacin or nitroimidazole derivatives such as metronidazole) that had not been on stable doses of these medications for at least 4 weeks prior to Baseline. In addition, subjects on aminosalicylates or Crohn's-related antibiotic treatments who had discontinued these medications within four weeks of Baseline.
23. Subjects on prednisone > 40 mg/day (or equivalent) or subjects on < 10 mg/day prednisone and subjects who were not on a stable dose for at least 2 weeks prior to Baseline. In addition, subjects who discontinued prednisone (or equivalent) within 2 weeks of Baseline.
24. Subjects on growth hormone that had not been on a stable dose for at least 12 weeks prior to Baseline. Subjects had to consent to remain on a stable dose through the duration of the study.
25. Subjects on budesonide > 9 mg/day and subjects who were not on stable doses for at least 2 weeks prior to Baseline. In addition, subjects who discontinued budesonide within 2 weeks of Baseline.
26. Subjects who were currently taking both budesonide and prednisone (or equivalent).
27. Subjects who had undergone therapeutic enemas within two weeks prior to Baseline.
28. Subjects who had been on cyclosporine (intravenous [IV], oral), tacrolimus (any form), or mycophenolate mofetil within 28 days of Baseline.
29. Subjects who had been on Kineret® (anakinra) must discontinue use 2 days prior to Baseline.
30. Subjects with any prior exposure to Tysabri (natalizumab).
31. Subjects with known hypersensitivity to the excipients of adalimumab as stated in the label.
32. Subjects with a previous history of dysplasia of the gastrointestinal tract.
33. Subjects who weighed < 17 kg at Screening.
34. Subject not in compliance with prior and concomitant medications.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Thakkar, Study Director — Abbott
Locations (45):
- United States (26):
  - Site Reference ID/Investigator# 10287, Los Angeles, California
  - Site Reference ID/Investigator# 5223, Orange, California
  - Site Reference ID/Investigator# 4984, San Francisco, California
  - Site Reference ID/Investigator# 5222, Aurora, Colorado
  - Site Reference ID/Investigator# 5676, Hartford, Connecticut
  - Site Reference ID/Investigator# 4911, Orlando, Florida
  - Site Reference ID/Investigator# 7640, Orlando, Florida
  - Site Reference ID/Investigator# 5904, Atlanta, Georgia
  - Site Reference ID/Investigator# 4316, Chicago, Illinois
  - Site Reference ID/Investigator# 5901, Maywood, Illinois
  - Site Reference ID/Investigator# 4912, Indianapolis, Indiana
  - Site Reference ID/Investigator# 4317, Baltimore, Maryland
  - Site Reference ID/Investigator# 5102, Rochester, Minnesota
  - Site Reference ID/Investigator# 4285, Saint Paul, Minnesota
  - Site Reference ID/Investigator# 3826, Las Vegas, Nevada
  - Site Reference ID/Investigator# 6182, Morristown, New Jersey
  - Site Reference ID/Investigator# 8801, Buffalo, New York
  - Site Reference ID/Investigator# 3734, Mineola, New York
  - Site Reference ID/Investigator# 4913, New Hyde Park, New York
  - Site Reference ID/Investigator# 6257, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 4909, Cincinnati, Ohio
  - Site Reference ID/Investigator# 4914, Columbus, Ohio
  - Site Reference ID/Investigator# 5892, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 6354, Nashville, Tennessee
  - Site Reference ID/Investigator# 4983, Seattle, Washington
  - Site Reference ID/Investigator# 4950, Milwaukee, Wisconsin
- Belgium (3):
  - Site Reference ID/Investigator# 6700, Antwerp
  - Site Reference ID/Investigator# 7744, Brussels
  - Site Reference ID/Investigator# 6073, Brussels
- Canada (7):
  - Site Reference ID/Investigator# 5109, Calgary
  - Site Reference ID/Investigator# 4916, Halifax
  - Site Reference ID/Investigator# 10284, Hamilton
  - Site Reference ID/Investigator# 8391, London
  - Site Reference ID/Investigator# 5169, Ottawa
  - Site Reference ID/Investigator# 6798, Toronto
  - Site Reference ID/Investigator# 5570, Vancouver
- Site Reference ID/Investigator# 6071, Prague, Czechia
- France (2):
  - Site Reference ID/Investigator# 6065, Paris
  - Site Reference ID/Investigator# 6072, Paris
- Netherlands (3):
  - Site Reference ID/Investigator# 16501, Amsterdam
  - Site Reference ID/Investigator# 14750, Nijmegen
  - Site Reference ID/Investigator# 13622, Rotterdam
- Poland (2):
  - Site Reference ID/Investigator# 6428, Warsaw
  - Site Reference ID/Investigator# 6430, Wroclaw
- Site Reference ID/Investigator# 7742, London, United Kingdom

REFERENCES:
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- [Derived] Ruemmele FM, Rosh J, Faubion WA, Dubinsky MC, Turner D, Lazar A, Eichner S, Maa JF, Alperovich G, Robinson AM, Hyams JS. Efficacy of Adalimumab for Treatment of Perianal Fistula in Children with Moderately to Severely Active Crohn's Disease: Results from IMAgINE 1 and IMAgINE 2. J Crohns Colitis. 2018 Nov 9;12(10):1249-1254. doi: 10.1093/ecco-jcc/jjy087. PMID 29939254
- [Derived] Hyams JS, Griffiths A, Markowitz J, Baldassano RN, Faubion WA Jr, Colletti RB, Dubinsky M, Kierkus J, Rosh J, Wang Y, Huang B, Bittle B, Marshall M, Lazar A. Safety and efficacy of adalimumab for moderate to severe Crohn's disease in children. Gastroenterology. 2012 Aug;143(2):365-74.e2. doi: 10.1053/j.gastro.2012.04.046. Epub 2012 May 2. PMID 22562021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 45 investigative sites in the US, Canada, and Europe. A total of 192 subjects received at least one dose of adalimumab and participated in the 4-week Open-label induction period of the study. Of these, 4 discontinued and 188 subjects participated in the DB Maintenance period.
Pre-assignment Details: Enrolled pediatric subjects were given an induction regimen of 160/80 mg adalimumab at Baseline/Week 2 or 80/40 mg at Baseline/Week 2 according to the subjects' Baseline body weight (BW) and were randomized at Week 4 to receive one of two maintenance regimens of adalimumab every other week (eow).
Groups:
- Open-label Adalimumab (Week 0 to Week 4): All subjects received an open-label adalimumab induction regimen. Subjects weighing ≥ 40 kg at Baseline received 160 mg at Week 0 and 80 mg at Week 2. Subjects weighing < 40 kg at Baseline received 80 mg at Week 0 and 40 mg at Week 2.
- Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52): Subjects randomized to the Low-Dose treatment group received either 20 mg adalimumab every other week (eow) (if Week 4 body weight [BW] ≥ 40 kg) or 10 mg adalimumab eow (if Week 4 BW < 40 kg). Starting at the Week 12 study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blind (DB) ew therapy they could be switched to open-label ew therapy.
- High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52): Subjects randomized to the High-Dose treatment group received either 40 mg adalimumab every other week (eow) (if Week 4 body weight [BW] ≥ 40 kg) or 20 mg adalimumab eow (if Week 4 BW < 40 kg). Starting at the Week 12 study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blinded (DB) ew therapy they could be switched to open-label ew therapy.
Period: Open-label Induction Period
Arm/Group | Open-label Adalimumab (Week 0 to Week 4) | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Started | 192 | 0 | 0
Completed | 188 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Subject did not satisfy entry criteria | 1 | 0 | 0
Period: EOW Double-blind Maintenance Period
Arm/Group | Open-label Adalimumab (Week 0 to Week 4) | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Started | 0 | 95 | 93
Completed | 0 | 58 | 66
Not Completed | 0 | 37 | 27
Not completed — Adverse Event | 0 | 10 | 12
Not completed — Lack of Efficacy | 0 | 18 | 11
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 4 | 1
Not completed — Non-compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52): Subjects randomized to the High-Dose treatment group received either 40 mg adalimumab every other week (eow) (if Week 4 body weight [BW] was greater than or equal to 40 kg) or 20 mg adalimumab eow (if Week 4 BW less than 40 kg). Starting at the Week 12study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blinded (DB) ew therapy they could be switched to open-label ew therapy.
- Low-Dose Adalimumab: 20 mg or 10 mg (Week 4 to Week 52): Subjects randomized to the Low-Dose treatment group received either 20 mg adalimumab every other week (eow) (if Week 4 body weight [BW] was greater than or equal to 40 kg) or 10 mg adalimumab eow (if Week 4 BW less than 40 kg). Starting at the Week 12study visit, subjects who experienced a disease flare or were non-responders could be switched from blinded eow dosing to blinded every week (ew) dosing, continuing with the same blinded dose. If a subject continued to experience a flare or met the definition of non-response following an 8-week course of double-blind (DB) ew therapy they could be switched to open-label ew therapy.
- Total: Total of all reporting groups
Arm/Group | Open-label Adalimumab (Week 0 to Week 4) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52) | Low-Dose Adalimumab: 20 mg or 10 mg (Week 4 to Week 52) | Total
Number analyzed (Participants) | 0 | 93 | 95 | 188
Age Continuous [Mean (Standard Deviation); unit: years] | 0 (0) | 13.7 (2.52) | 13.5 (2.47) | 13.6 (2.49)
Age, Customized [Number; unit: years]
  < 13 | 0 | 31 | 35 | 66
  >= 13 | 0 | 62 | 60 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 42 | 41 | 83
  Male | 0 | 51 | 54 | 105
Race/Ethnicity, Customized [Number; unit: participants]
  White | 0 | 81 | 85 | 166
  Black | 0 | 5 | 6 | 11
  Asian | 0 | 3 | 0 | 3
  American Indian/Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Mult-race | 0 | 1 | 2 | 3
  Other | 0 | 3 | 2 | 5
Weight [Number; unit: kg]
  < 40 | 0 | 32 | 35 | 67
  >= 40 | 0 | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Clinical Remission as Defined by Pediatric Crohn's Disease Activity Index (PCDAI) Score ≤ 10 at Week 26
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. The primary endpoint was clinical remission as defined by PCDAI score ≤ 10. The comparison was between High-Dose adalimumab versus Low-Dose adalimumab in the intent-to-treat population.
Time Frame: Week 26
Population: Comparison of adalimumab High-Dose versus Low-Dose with respect to the primary efficacy endpoint in the intent-to-treat analysis set as all randomized subjects who received at least one dose of double-blind study medication.
Measure: Number; unit: percent of participants
Arm/Group | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Number analyzed (Participants) | 95 | 93
percent of participants | 28.4 | 38.7
Statistical Analysis 1: Comparison: Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) vs High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52); The point estimates for the number of subjects who achieved PCDAI clinical remission in each treatment group and the difference in number between the groups were provided. The P value and 95% confidence intervals (CIs) for the difference were provided. The P value is from the CMH test adjusted for infliximab use and response status at Week 4. The primary analysis was performed for the intent-to-treat (ITT) using the non-responder (NRI) imputation method; Test type: Superiority or Other; p = 0.075, Cochran-Mantel-Haenszel — There is no adjustment for multiple comparison on the primary outcome measure; Mean Difference (Net) = 10.29, 95% CI 2-sided [-3.14 to 23.71] — Difference is between adalimumab High-dose and adalimumab Low-dose group

2. Secondary Outcome: Percent of Participants With Clinical Remission as Defined by Pediatric Crohn's Disease Activity Index (PCDAI) Score ≤ 10 at Week 52
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit erythrocyte sedimentation rate, albumin, weight, height, examination of abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100 with higher scores indicating more active disease. Clinical remission was defined as PCDAI score of ≤ 10.
  The comparison was between High-Dose adalimumab versus Low-Dose adalimumab in the intent-to treat population.
Time Frame: Week 52
Population: Intent-to-treat population using non-responder imputation method.
Measure: Number; unit: percent of participants
Arm/Group | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Number analyzed (Participants) | 95 | 93
percent of participants | 23.2 | 33.3
Statistical Analysis 1: Comparison: Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) vs High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52); The point estimates for the number of subjects who achieved PCDAI clinical remission in each treatment group and the difference in number between the groups were provided. The P value and 95% CIs for the difference were provided. The analysis was performed for the intent-to-treat (ITT) population using the non-responder imputation (NRI) method; Test type: Superiority or Other; p = 0.100, Cochran-Mantel-Haenszel — The hierarchical stepwise closed testing procedure was implemented to control the overall significance level at 0.05 in the ITT population; Mean Difference (Net) = 10.18, 95% CI 2-sided [-2.62 to 22.97] — A significance test for any individual major secondary efficacy endpoint in the hierarchy was to be inferential only if the hypothesis tests of all preceding major secondary efficacy endpoints were statistically significant at 0.050

3. Secondary Outcome: Percent of Participants With Clinical Response as Defined by Pediatric Crohn's Disease Activity Index (PCDAI) Score at Week 26
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, examination of abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical response was defined as a decrease from Baseline in the PCDAI score of at least 15 points. The comparison was High-Dose adalimumab versus Low-Dose in the ITT population.
Time Frame: Week 26
Population: Intent-to-treat population using non-responder imputation (NRI) method.
Measure: Number; unit: percent of participants
Arm/Group | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Number analyzed (Participants) | 95 | 93
percent of participants | 48.4 | 59.1
Statistical Analysis 1: Comparison: Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) vs High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52); The point estimates for the number of subjects who achieved PCDAI clinical response in each treatment group and the difference in number between the groups were provided. The P value and 95% confidence intervals (CIs) for the difference were provided. The analysis was performed for the intent-to-treat (ITT) population using the non-responder imputation (NRI) method; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 10.72, 95% CI 2-sided [-3.45 to 24.89] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percent of Participants With Clinical Response as Defined by Pediatric Crohn's Disease Activity Index (PCDAI) Score at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: Intent-to-treat population using non-responder imputation (NRI) method.
Measure: Number; unit: percent of participants
Arm/Group | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Number analyzed (Participants) | 95 | 93
percent of participants | 28.4 | 41.9
Statistical Analysis 1: Comparison: Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) vs High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.038, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 13.51, 95% CI 2-sided [-0.01 to 27.04] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline IMPACT III Scores at Week 26 (Observed Case)
Description: The IMPACT III questionnaire is a 35-item assessment of health-related quality of life in patients with inflammatory bowel disease (Crohn's disease [CD] or ulcerative colitis). In this study, subjects greater than or equal 10 years old who had CD at baseline completed an IMPACT III questionnaire at Baseline, Week 26, and Week 52. Subjects marked an option from 1 to 5 for each item left to right with numbers 5 (good 'quality of life' condition) through 1 (bad 'quality of life' condition). The total scores, range from 35 to 175 with higher scores representing a better quality of life.
Time Frame: Baseline and Week 26
Population: Intent-to-treat (ITT) population for observed case (OC).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Number analyzed (Participants) | 48 | 56
Scores on a scale | 26.40 (15.589) | 23.70 (18.990)
Statistical Analysis 1: Comparison: Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) vs High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52); Analyzed as change from Baseline to Week 26, and compared between the two treatment groups. The estimated treatment mean difference, P values, and 95% CI for the treatment difference were provided. Analysis was conducted in the ITT population for OC. The P value is from the ANCOVA model with treatment as a factor, adjusted for the baseline value, and the strata (response status at Week 4 and prior infliximab experience); Test type: Superiority or Other; p = 0.161, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.10, 95% CI 2-sided [-9.86 to 1.66], Standard Error of Mean 2.903 — Difference is between adalimumab High-dose and adalimumab Low-dose groups. Baseline means include subjects who had both Baseline and post-Baseline measurements

6. Secondary Outcome: Change From Baseline IMPACT III Scores at Week 52 (Observed Case)
Description: as for outcome 5
Time Frame: Baseline and Week 52
Population: Intent-to-treat (ITT) population for observed case (OC).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Number analyzed (Participants) | 31 | 38
Scores on a scale | 26.49 (16.182) | 24.25 (14.678)
Statistical Analysis 1: Comparison: Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) vs High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52); Analyzed as change from Baseline to Week 52, and compared between the two treatment groups. The estimated treatment mean difference, P values, and 95% confidence interval (CI) for the treatment difference were provided. Analysis was conducted in the ITT population for OC; Test type: Superiority or Other; p = 0.735, ANCOVA; Mean Difference (Net) = -1.00, 95% CI 2-sided [-6.88 to 4.88], Standard Error of Mean 2.941 — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) reported from the time of study drug administration until 70 days after discontinuation of study drug were collected. Serious AEs were collected from the time the subject or parent/legal guardian signed the informed consent.
Description: Open-label (OL) Adalimumab (Wk 0 - Wk 4): AEs from first OL dose to 70 days after last OL induction adalimumab dose or until first double-blind (DB) dose Low-Dose/High-Dose Adalimumab (Wk 4 - Wk 52): AEs from first DB dose to 70 days after last DB every other week (eow) or until switch to every week (ew) dosing or OL extension
Arm/Group | Open-label Adalimumab (Week 0 to Week 4) | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52)
Serious Adverse Events (participants affected / at risk) | 6/192 | 19/95 | 22/93
Other Adverse Events (participants affected / at risk) | 64/192 | 62/95 | 69/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Adalimumab (Week 0 to Week 4) (N=192) | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) (N=95) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52) (N=93)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 4
CROHN'S DISEASE (Gastrointestinal disorders) | 2 | 15 | 12
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 1
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 1
BARTHOLIN'S ABSCESS (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
H1N1 INFLUENZA (Infections and infestations) | 0 | 0 | 1
HISTOPLASMOSIS DISSEMINATED (Infections and infestations) | 0 | 0 | 1
SCARLET FEVER (Infections and infestations) | 0 | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0
YERSINIA INFECTION (Infections and infestations) | 1 | 0 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
HEART RATE IRREGULAR (Investigations) | 1 | 0 | 0
PSYCHOSOMATIC DISEASE (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Adalimumab (Week 0 to Week 4) (N=192) | Low-Dose Adalimumab: 20 mg or 10 mg Eow (Week 4 to Week 52) (N=95) | High-Dose Adalimumab: 40 mg or 20 mg Eow (Week 4 to Week 52) (N=93)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 6 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 6 | 9
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 3 | 7
CROHN'S DISEASE (Gastrointestinal disorders) | 5 | 15 | 11
DIARRHOEA (Gastrointestinal disorders) | 3 | 9 | 8
NAUSEA (Gastrointestinal disorders) | 9 | 6 | 10
VOMITING (Gastrointestinal disorders) | 3 | 10 | 6
FATIGUE (General disorders) | 3 | 4 | 5
INJECTION SITE PAIN (General disorders) | 12 | 4 | 2
INJECTION SITE REACTION (General disorders) | 10 | 4 | 5
PAIN (General disorders) | 2 | 2 | 5
PYREXIA (General disorders) | 1 | 8 | 10
NASOPHARYNGITIS (Infections and infestations) | 3 | 11 | 9
PHARYNGITIS (Infections and infestations) | 2 | 2 | 7
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 5 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 10 | 10
VIRAL INFECTION (Infections and infestations) | 0 | 6 | 4
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 3 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 5 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 5
DIZZINESS (Nervous system disorders) | 2 | 5 | 1
HEADACHE (Nervous system disorders) | 9 | 20 | 16
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 9
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 9
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 3
RASH (Skin and subcutaneous tissue disorders) | 0 | 5 | 5

LIMITATIONS AND CAVEATS:
Absence of placebo group comparative data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.